CLINICAL TRIAL: NCT06528964
Title: Expression of Proteinopathies in Skin Biopsies of Patients With Neurodegenerative Disorders
Brief Title: Proteinopathies Expression in Skin of Neurodegenerative Disorders
Status: Recruiting | Type: Observational
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Ildefonso Rodriguez-Leyva, Head of Neurology Service, Universidad Autonoma de San Luis Potosí
Other Study IDs: 42-23
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease; Frontotemporal Dementia; Parkinson Disease; Atypical Parkinsonism; Amyotrophic Lateral Sclerosis; Normal Pressure Hydrocephalus
Keywords: Alpha Synuclein Pathology; Tauopathies; TDP-43 Proteinopathies; Beta-Amyloid
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Parkinson Disease; Amyotrophic Lateral Sclerosis; Hydrocephalus, Normal Pressure; Synucleinopathies; Tauopathies; TDP-43 Proteinopathies; Plaque, Amyloid | interventions — Immunohistochemistry; Fluorescent Antibody Technique

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 4mm skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with neurodegenerative disease: Patients diagnosed with either Alzheimer's disease, frontotemporal lobe dementia, Parkinson's disease, atypical Parkinsonism or amyotrophic lateral sclerosis.
  Interventions: Diagnostic Test: Immunohistochemistry and immunofluorescence
- Patients with normal pressure hydrocephalus: Patients diagnosed with normal pressure hydrocephalus, because of their clinical presentation (acute or subacute gait abnormalities, memory loss or personality changes and urinary incontinence) with radiological confirmation of ventriculomegaly and normal cerebrospinal fluid opening pressure.
  Interventions: Diagnostic Test: Immunohistochemistry and immunofluorescence
- Healthy control subjects: Person, men or women, above 45 years old, that don't have history of family or personal neurodegenerative disease.
  Interventions: Diagnostic Test: Immunohistochemistry and immunofluorescence

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry and immunofluorescence — Skin biopsies will be analyzed using immunohistochemistry and immunofluorescence to detect the presence of aggregated a-synuclein, amyloid-b, p-TAU and TDP-43.

SUMMARY:
The goal of this observational study is to compare the aggregation pattern of proteinopathies (alpha-synuclein, amyloid-beta, phosphorylated tau and transactive response DNA -binding protein 43 [TDP43]) in skin biopsies of patients with a neurodegenerative disease like Alzheimer's disease, frontotemporal lobe dementia, Parkinson's disease, atypical Parkinsonism, amyotrophic lateral sclerosis or normal pressure hydrocephalus. The main question it aims to answer is:

* Is there a specific pattern of aggregation of proteinopathies in skin biopsies in each neurodegenerative disease in comparison to healthy control subjects?

Skin biopsies will be analyzed using immunohistochemistry and immunofluorescence for detection of alpha-synuclein, amyloid-beta, phosphorylated tau and TAR DNA binding protein 43, and the aggregation patterns will be compared between patients with a neurodegenerative disease vs patient with normal pressure hydrocephalus vs healthy control subjects.

DETAILED DESCRIPTION:
Alzheimer's disease is the main cause of neurodegenerative dementia and represents a high degree of morbidity and mortality among the patients who have it, causing a great economic impact in health systems. In general population the second cause of neurodegenerative dementia is frontotemporal lobe dementia and it's also the first cause of dementia in patients under 65 years old.

Neurodegenerative diseases have been associated with the deposit of abnormal aggregated proteins like alpha-synuclein, amyloid-beta, phosphorylated tau and TAR DNA binding protein 43 in brain tissue. Similar deposits of a-synuclein, p-TAU and TDP-43 have been identified through immunohistochemistry and immunofluorescence in skin biopsies.

Main objective: Compare the aggregation pattern between the different proteinopathies (a-synuclein, amyloid-b, p-TAU and TDP-43) with immunohistochemistry in skin biopsies of patients with Alzheimer's disease, frontotemporal lobe dementia, Parkinson's disease, atypical Parkinsonism, amyotrophic lateral sclerosis and normal pressure hydrocephalus vs control subjects.

Study design: this will be an observational, transversal and comparative analysis study. Inclusion criteria: patients, men and women, 45 and older diagnosed with Alzheimer's disease, frontotemporal lobe dementia, Parkinson's disease, atypical Parkinsonism, amyotrophic lateral sclerosis or normal pressure hydrocephalus will be recruited for sampling with skin biopsy. Healthy control subjects will be men or women similar in age to the patients that don't have any personal or family history of a neurodegenerative disease and that are not related by blood to the patients in this study.

Sample size calculation and statistical analysis:

All the patients that meet the inclusion criteria and accept the consent form, from the neurology department of Hospital Central Dr Ignacio Morones Prieto, will be recruited for one year.

A descriptive analysis will be carried out with frequencies and percentages for categorical variables, for continuous variables central tendency and dispersion analysis, the normality of the data will be evaluated using the Kolmogorov-Smirnov or Shapiro-Wilk test as appropriate. In case the data ha a normal distribution, it will be analyzed with the ANOVA test followed by Tukey and in the case the data doesn't have a normal distribution the analysis will be made with Kruskal Wallis followed by Mann Whitney U.

ELIGIBILITY:
Inclusion Criteria for patients:

* Patients 45 years and older
* Men and women
* Patients diagnosed with Alzheimer's disease, frontotemporal lobe dementia, Parkinson's disease, atypical Parkinsonism, amyotrophic lateral sclerosis or normal pressure hydrocephalus
* Patients that voluntarily accept to participate in the study and accept the consent form

Inclusion Criteria healthy control subjects:

* People 45 years and older
* Men and women
* Subjects can be related to a patient but not by blood (for example spouse of a patient)
* Subjects don't have direct family history of a neurodegenerative control
* Subjects don't have any clinical findings suggesting dementia
* Subjects voluntarily accept to participate in the study and accept the consent form

Exclusion Criteria:

* Patients or controls that have a personal history of cerebrovascular disease, psychiatric disease, post traumatic dementia or HIV related dementia
* Patients in which the diagnosis is not clear or hasn't been confirmed
* Patients or controls that have a neuroinfection
* Patients or controls that a diagnosed skin disease
* Patients that have an "atypical" presentation of the disease
* Patients or controls that have diagnosis of a coagulopathy

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients and controls that meet the eligibility criteria will be recruited from the neurology department consult from the Hospital Central Dr Ignacio Morones Prieto
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Aggregation pattern of a-synuclein, amyloid-b, p-TAU and TDP-43 | Each patient will be recruited and sampled the same day of the evaluation which will take about 1 hour. The final report it takes a frame time around two years.
  The detection of each proteinopathy will be compared between each of them in every patient and compared to healthy control subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Said HM, Kaya D, Yavuz I, Dost FS, Altun ZS, Isik AT. A Comparison of Cerebrospinal Fluid Beta-Amyloid and Tau in Idiopathic Normal Pressure Hydrocephalus and Neurodegenerative Dementias. Clin Interv Aging. 2022 Apr 11;17:467-477. doi: 10.2147/CIA.S360736. eCollection 2022. PMID 35431542
- [Background] Espay AJ, Da Prat GA, Dwivedi AK, Rodriguez-Porcel F, Vaughan JE, Rosso M, Devoto JL, Duker AP, Masellis M, Smith CD, Mandybur GT, Merola A, Lang AE. Deconstructing normal pressure hydrocephalus: Ventriculomegaly as early sign of neurodegeneration. Ann Neurol. 2017 Oct;82(4):503-513. doi: 10.1002/ana.25046. Epub 2017 Oct 4. PMID 28892572
- [Background] Castanedo-Cazares JP, Rodriguez-Leyva I. Skin biomarkers for neurodegenerative disease: a future perspective. Neurodegener Dis Manag. 2015 Dec;5(6):465-7. doi: 10.2217/nmt.15.51. Epub 2015 Nov 30. No abstract available. PMID 26619251
- [Background] Rodriguez-Leyva I, Chi-Ahumada EG, Carrizales J, Rodriguez-Violante M, Velazquez-Osuna S, Medina-Mier V, Martel-Gallegos MG, Zarazua S, Enriquez-Macias L, Castro A, Calderon-Garciduenas AL, Jimenez-Capdeville ME. Parkinson disease and progressive supranuclear palsy: protein expression in skin. Ann Clin Transl Neurol. 2016 Feb 1;3(3):191-9. doi: 10.1002/acn3.285. eCollection 2016 Mar. PMID 27042679
- [Background] Golde TE, Borchelt DR, Giasson BI, Lewis J. Thinking laterally about neurodegenerative proteinopathies. J Clin Invest. 2013 May;123(5):1847-55. doi: 10.1172/JCI66029. Epub 2013 May 1. PMID 23635781